CLINICAL TRIAL: NCT01520506
Title: Rapid Renal Sympathetic Denervation for Resistant Hypertension Using the OneShot™ Ablation System
Brief Title: Rapid Renal Sympathetic Denervation for Resistant Hypertension
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: Medtronic - MITG (Industry); Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 012
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Hypertension; Kidney Diseases; Kidney Failure, Chronic; Vascular Diseases; Cardiovascular Diseases; Urologic Diseases; Renal Insufficiency, Chronic; Renal Insufficiency
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Hypertension; Kidney Diseases; Kidney Failure, Chronic; Vascular Diseases; Cardiovascular Diseases; Urologic Diseases; Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapid Renal Denervation (Experimental)
  Interventions: Device: Covidien OneShot™ System

INTERVENTIONS:
Device: Covidien OneShot™ System — Placed percutaneously, the OneShot™ balloon catheter is advanced into the renal artery using a routine femoral approach in a cardiac catheterization laboratory setting. RF is applied with pre-programmed time and intensity in each of the renal arteries.
  Other Names: Covidien OneShot™ Renal Denervation System

SUMMARY:
The Covidien OneShot™ ablation system use is to deliver low-level radio frequency (RF) energy through the wall of the renal artery to denervate the human kidney.

DETAILED DESCRIPTION:
Unique to the OneShot™ ablation system is the ability to deliver the desired helical treatment pattern for optimal Renal Denervation (RDN) with a single balloon based-treatment, eliminating user variance inherent in the currently available point-by-point approach. In addition, technological improvements have been incorporated. The OneShot™ RF generator has a touchscreen, user friendly interface; catheter advancement is made safer with the use of a guidewire; two radiopaque markers on the catheter enable more precise device positioning; and the irrigated catheter tip reduces the risk of overheating and clot formation during RF delivery. By offering a more reliable single treatment approach, coupled with enhanced ease-of use and reduced procedure times, this technology has the potential to significantly expand clinical adoption of catheter-based renal sympathetic denervation.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic blood pressure ≥ 160 mmHg despite treatment with a regimen of 3 or more anti-hypertensive medications that includes a diuretic and that has been stable for 2 weeks prior to screening.
2. Age 18-85 years.
3. Able to provide informed consent and comply with follow-up visits.

Exclusion Criteria:

1. Diameter of left or right renal artery less than 4 mm or greater than 7mm.
2. Length of target segment of left or right renal artery less than 20mm.
3. Other renal arterial abnormalities including severe renal artery stenosis, previous renal stenting or angioplasty.
4. End-stage renal disease requiring dialysis or renal transplant.
5. estimated Glomerular Filtration Rate < 45 mL/min per 1.73 m2.
6. Type 1 diabetes mellitus.
7. Myocardial infarction, unstable angina, or cerebrovascular events within 6 months prior to screening.
8. Severe valvular heart disease for which reduction of blood pressure would be considered hazardous.
9. Bleeding disorder or refusing blood transfusions.
10. Pregnancy or breast feeding.
11. Peripheral vascular disease precluding catheter insertion.
12. Any serious medical condition, which in the opinion of the investigator, may adversely affect the safety or effectiveness of the participant or the study.
13. Current enrollment in another investigational drug or device Study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W.A.L. Tonino, MD, Principal Investigator — Department of Cardiology, Catherina Hospital, Eindhoven, The Netherlands; Stefan Verheye, MD, Principal Investigator — Department of Interventional Cardiology, Middelheim Hospital, Antwerp, Belgium
Locations (14):
- Belgium (2):
  - Middelheim Hospital, Antwerp
  - Ziekenhuis Oost--Limburg, Genk
- Germany (5):
  - Universitatklinikum, Bonn
  - Cardiovascular Center Sankt Katharinen, Frankfurt
  - Asklepios Klinik St. Georg, Hamburg
  - Univ. Medical Klinik III, Heidelberg
  - Franziskus Hospital, Münster
- Hospital San Raffaele, Milan, Italy
- Centre Hospitalier De Luxembourg, Luxembourg, Luxembourg
- Netherlands (4):
  - Santa Catharina Hospital, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC Thoraxcenter, Rotterdam
  - UMC Universitair Medisch Centrum, Utrecht
- Mercy Angiography Unit, Auckland, New Zealand

REFERENCES:
- [Derived] Verheye S, Ormiston J, Bergmann MW, Sievert H, Schwindt A, Werner N, Vogel B, Colombo A. Twelve-month results of the rapid renal sympathetic denervation for resistant hypertension using the OneShotTM ablation system (RAPID) study. EuroIntervention. 2015 Feb;10(10):1221-9. doi: 10.4244/EIJY14M12_02. PMID 25452198
- See also: Covidien (manufacturer) — http://www.covidien.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapid Renal Denervation: Covidien OneShot™ System: Placed percutaneously, the OneShot™ balloon catheter is advanced into the renal artery using a routine femoral approach in a cardiac catheterization laboratory setting. Radiofrequency (RF) is applied with pre-programmed time and intensity in each of the renal arteries.
Period: Overall Study
Arm/Group | Rapid Renal Denervation
Started | 50
Completed | 44
Not Completed | 6
Not completed — Missed Visit | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rapid Renal Denervation
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Acute Procedural Safety
Description: Acute Procedural Safety, defined as the overall rate of Serious Adverse Events (SAE's) and adverse device effects at discharge:
  * SAE's related to groin and vascular access complications, and
  * SAE's related to renal artery injury.
Time Frame: One Week
Measure: Number; unit: percentage of participants
Arm/Group | Rapid Renal Denervation
Number analyzed (Participants) | 50
percentage of participants | 4

2. Secondary Outcome: Chronic Procedural Safety
Description: Chronic Procedural Safety, defined as the overall rate of Serious Adverse Events and Adverse Device Effects at 6 months
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Rapid Renal Denervation
Number analyzed (Participants) | 50
percentage of participants | 6

3. Secondary Outcome: Renal Denervation Procedure Effectiveness
Description: Procedural Effectiveness, defined as rate of Office Systolic Blood Pressure (SBP) reduction > 10 mmHg at 6 months compared to baseline
Time Frame: From baseline to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Rapid Renal Denervation
Number analyzed (Participants) | 47
percentage of participants | 61.7

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rapid Renal Denervation
Serious Adverse Events (participants affected / at risk) | 16/50
Other Adverse Events (participants affected / at risk) | 32/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Renal Denervation (N=50)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders (Cardiac disorders) | 7 (8)
General disorders and administrative site conditions (General disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)
Vascular disorders (Vascular disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Renal Denervation (N=50)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorders (Cardiac disorders) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3)
General disorders and administrative site conditions (General disorders) | 7 (7)
Infections and infestations (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3)
Investigations (Investigations) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3)
Nervous system disorders (Nervous system disorders) | 7 (7)
Psychiatric disorders (Psychiatric disorders) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Vascular disorders (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results without permission of the sponsor.